CLINICAL TRIAL: NCT01751698
Title: Adaptive Interventions for Minimally Verbal Children With ASD in the Community
Acronym: AIM-ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD073975 (NIH); R01HD073975 (NIH)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Autism
Keywords: Autism; Minimally Verbal; School Age
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JASP-EMT (Active Comparator): JASP-EMT (Joint Attention, Symbolic Play and Enhanced Milieu Teaching) focuses on creating a context for joint engagement within naturally occurring child-led play routines. There is evidence of the effects of these interventions with children with ASD, and pilot data showing effects with minimally verbal children.
  Interventions: Behavioral: JASP-EMT
- DTT (Active Comparator): CORE-DTT (discrete trial training for core features of ASD) emphasizes didactic adult-led instruction and is considered the current evidenced-based 'standard of care' for children with autism (NRC, 2001).
  Interventions: Behavioral: DTT

INTERVENTIONS:
Behavioral: JASP-EMT — JASP-EMT is a developmentally anchored behavioral intervention that assumes that communication develops from social interactions in which specific social engagement strategies, symbolic representations, and early communication forms are modeled and naturally reinforced by adult partner responses to the child. The goal of JASP-EMT is to increase (a) joint engagement, (b) initiating joint attention gestures, (c) social play involving objects and persons, and (d) verbal and nonverbal communication by facilitating meaningful social interactions. The social interaction foundation of JASP-EMT is critical. Modeling and expansions of communicative behaviors and play are used strategically within meaningful social interactions with therapists and caregivers.
  Arms: JASP-EMT
Behavioral: DTT — CORE-DTT is based on behavioral learning theory in which communication and related skills are taught through systematic direct instruction. The goal of CORE-DTT is to help children be successful in learning communication skills by breaking these skills down into small steps, providing systematic direct instruction on each step, and reinforcing children (e.g., with praise or access to preferred items) for demonstrating skills. Imitation and attention skills are a main focus early in intervention. DTT is the most common evidence-based approach for teaching children with ASD, and is often considered the closest to a 'standard of practice' for the field.
  Arms: DTT

SUMMARY:
Adaptive Interventions for Minimally Verbal Children with ASD in the Community, seeks support to construct an adaptive intervention that utilizes two efficacious interventions (JASP-EMT and CORE- DTT) that have shown promise for optimizing the number of unique socially communicative and spontaneously spoken words in minimally verbal children with ASD. The study utilizes a novel sequential multiple assignment-randomized trial to evaluate and construct an optimal adaptive intervention. A total of 192 minimally verbal school aged children with an Autism Spectrum Disorder (aged 5 to 8 years of age) will participate across four sites, University of California Los Angeles, University of Rochester, Vanderbilt University and Weill Cornell Medical Center with methodological and statistical support from University of Michigan.

DETAILED DESCRIPTION:
Interventions:

* CORE-DTT is based on behavioral learning theory in which communication and related skills are taught through systematic direct instruction. The goal of CORE-DTT is to help children be successful in learning communication skills by breaking these skills down into small steps, providing systematic direct instruction on each step, and reinforcing children (e.g., with praise or access to preferred items) for demonstrating skills. Imitation and attention skills are a main focus early in intervention. DTT is the most common evidence-based approach for teaching children with ASD, and is often considered the closest to a 'standard of practice' for the field. The participants in the proposed study will have had at least 1 year of previous intervention, likely in an ABA program with DTT as a main strategy. While many children will have been exposed to DTT prior to entering this trial, it is important to insure that children (a) receive quality DTT, and (b) have exposure to CORE elements related to language learning, specifically joint attention and requesting gestures, in order to make the comparison with JASP-EMT.
* JASP-EMT is a developmentally anchored behavioral intervention that assumes that communication develops from social interactions in which specific social engagement strategies, symbolic representations, and early communication forms are modeled and naturally reinforced by adult partner responses to the child. The goal of JASP-EMT is to increase (a) joint engagement, (b) initiating joint attention gestures, (c) social play involving objects and persons, and (d) verbal and nonverbal communication by facilitating meaningful social interactions. The social interaction foundation of JASP-EMT is critical. Modeling and expansions of communicative behaviors and play are used strategically within meaningful social interactions with therapists and caregivers. For minimally verbal children with autism, meaningful social interaction is essential for establishing the platform on which language input and development will be built.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism
* At least 4 years, 6 months old, and not older than 8 years, 0 months
* Displays less than 20 spontaneous, unique, and socially communicative words during screening assessments
* At least 18 months developmental age
* Currently in school

Exclusion Criteria:

* Diagnosis of syndrome or degenerative disorder
* Poorly controlled seizures

Ages: 54 Months to 96 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Primary Outcome 1: Language Sample | Follow-Up; 8 months on average
  To determine which intervention for minimally verbal children (JASP-EMT vs. CORE-DTT) produces greater increases in socially communicative spontaneous utterances (SCU; primary outcome).

SECONDARY OUTCOMES:
Secondary Aim 1: Joint Engagement | Follow-Up; 8 months on average
  To determine which intervention for minimally verbal children (JASP-EMT vs. CORE-DTT) produces greater increases in symbol-infused joint engagement.
Secondary Outcome 2: Number of Unique Words (Vocabulary) | Follow-Up; 8 months on average
  To determine which intervention for minimally verbal children (JASP-EMT vs. CORE-DTT) produces greater increases in number of unique words.
Secondary Outcome 3: Object Play | Follow-Up; 8 months on average
  To determine which intervention for minimally verbal children (JASP-EMT vs. CORE-DTT) produces greater increases in object play level.

OTHER OUTCOMES:
Parent Training | Follow-Up; 8 months on average
  To determine whether adding a parent training component provides additional benefit among participants who demonstrate a positive early response to either JASP-EMT or CORE-DTT.
Treatment Effects | Follow-Up; 8 months on average
  To compare and contrast four pre-specified adaptive interventions in terms of primary and secondary outcomes.
Moderators | Follow-Up; 8 months on average
  To determine whether (a) baseline repetitive behavior, (b) baseline object interest, and (c) parent expectations for the specific intervention moderate intervention outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, PhD, Principal Investigator — University of California, Los Angeles; Ann Kaiser, PhD, Principal Investigator — Vanderbilt University; Tristram Smith, PhD, Principal Investigator — University of Rochester; Catherine Lord, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - University of Rochester, Rochester, New York
  - Weill Cornell Medical College, White Plains, New York
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Kasari C, Paparella T, Freeman S, Jahromi LB. Language outcome in autism: randomized comparison of joint attention and play interventions. J Consult Clin Psychol. 2008 Feb;76(1):125-37. doi: 10.1037/0022-006X.76.1.125. PMID 18229990
- [Background] Kasari C, Freeman S, Paparella T. Joint attention and symbolic play in young children with autism: a randomized controlled intervention study. J Child Psychol Psychiatry. 2006 Jun;47(6):611-20. doi: 10.1111/j.1469-7610.2005.01567.x. PMID 16712638
- [Background] Kaiser AP, Roberts MY. Parent-implemented enhanced milieu teaching with preschool children who have intellectual disabilities. J Speech Lang Hear Res. 2013 Feb;56(1):295-309. doi: 10.1044/1092-4388(2012/11-0231). Epub 2012 Jun 28. PMID 22744141
- [Background] Roberts MY, Kaiser AP. Assessing the effects of a parent-implemented language intervention for children with language impairments using empirical benchmarks: a pilot study. J Speech Lang Hear Res. 2012 Dec;55(6):1655-70. doi: 10.1044/1092-4388(2012/11-0236). Epub 2012 Apr 5. PMID 22490620
- [Background] Smith T, Scahill L, Dawson G, Guthrie D, Lord C, Odom S, Rogers S, Wagner A. Designing research studies on psychosocial interventions in autism. J Autism Dev Disord. 2007 Feb;37(2):354-66. doi: 10.1007/s10803-006-0173-3. PMID 16897380
- [Background] Lord C, Wagner A, Rogers S, Szatmari P, Aman M, Charman T, Dawson G, Durand VM, Grossman L, Guthrie D, Harris S, Kasari C, Marcus L, Murphy S, Odom S, Pickles A, Scahill L, Shaw E, Siegel B, Sigman M, Stone W, Smith T, Yoder P. Challenges in evaluating psychosocial interventions for Autistic Spectrum Disorders. J Autism Dev Disord. 2005 Dec;35(6):695-708; discussion 709-11. doi: 10.1007/s10803-005-0017-6. PMID 16496206
- [Background] Pickett E, Pullara O, O'Grady J, Gordon B. Speech acquisition in older nonverbal individuals with autism: a review of features, methods, and prognosis. Cogn Behav Neurol. 2009 Mar;22(1):1-21. doi: 10.1097/WNN.0b013e318190d185. PMID 19372766
- [Background] Kidwell KM, Seewald NJ, Tran Q, Kasari C, Almirall D. Design and Analysis Considerations for Comparing Dynamic Treatment Regimens with Binary Outcomes from Sequential Multiple Assignment Randomized Trials. J Appl Stat. 2018;45:1628-1651. doi: 10.1080/02664763.2017.1386773. Epub 2017 Oct 12. PMID 30555200
- [Background] Almirall D, Kasari C, McCaffrey DF, Nahum-Shani I. Developing Optimized Adaptive Interventions in Education. J Res Educ Eff. 2018;11(1):27-34. doi: 10.1080/19345747.2017.1407136. Epub 2017 Nov 29. PMID 29552270
- [Background] Lu X, Nahum-Shani I, Kasari C, Lynch KG, Oslin DW, Pelham WE, Fabiano G, Almirall D. Comparing dynamic treatment regimes using repeated-measures outcomes: modeling considerations in SMART studies. Stat Med. 2016 May 10;35(10):1595-615. doi: 10.1002/sim.6819. Epub 2015 Dec 6. PMID 26638988
- [Background] Kasari C. Update on behavioral interventions for autism and developmental disabilities. Curr Opin Neurol. 2015 Apr;28(2):124-9. doi: 10.1097/WCO.0000000000000185. PMID 25695136
- [Result] Kasari C, Shire S, Shih W, Landa R, Levato L, Smith T. Spoken language outcomes in limited language preschoolers with autism and global developmental delay: RCT of early intervention approaches. Autism Res. 2023 Jun;16(6):1236-1246. doi: 10.1002/aur.2932. Epub 2023 Apr 18. PMID 37070270
- [Result] Sterrett K, Holbrook A, Landa R, Kaiser A, Kasari C. The effect of responsiveness to speech-generating device input on spoken language in children with autism spectrum disorder who are minimally verbaldagger. Augment Altern Commun. 2023 Mar;39(1):23-32. doi: 10.1080/07434618.2022.2120070. Epub 2022 Oct 20. PMID 36267016
- [Result] Toolan C, Holbrook A, Schlink A, Shire S, Brady N, Kasari C. Using the Clinical Global Impression scale to assess social communication change in minimally verbal children with autism spectrum disorder. Autism Res. 2022 Feb;15(2):284-295. doi: 10.1002/aur.2638. Epub 2021 Nov 19. PMID 34800004
- [Result] Harrop C, Sterrett K, Shih W, Landa R, Kaiser A, Kasari C. Short-term trajectories of restricted and repetitive behaviors in minimally verbal children with autism spectrum disorder. Autism Res. 2021 Aug;14(8):1789-1799. doi: 10.1002/aur.2528. Epub 2021 May 7. PMID 33960125
- [Result] Harrop C, Tu N, Landa R, Kasier A, Kasari C. Sensory Behaviors in Minimally Verbal Children With Autism Spectrum Disorder: How and When Do Caregivers Respond? Am J Intellect Dev Disabil. 2018 Jan;123(1):1-16. doi: 10.1352/1944-7558-123.1.1. PMID 29281320
- [Result] Kasari C, Sturm A, Shih W. SMARTer Approach to Personalizing Intervention for Children With Autism Spectrum Disorder. J Speech Lang Hear Res. 2018 Nov 8;61(11):2629-2640. doi: 10.1044/2018_JSLHR-L-RSAUT-18-0029. PMID 30418492
- [Result] Chang YC, Shih W, Landa R, Kaiser A, Kasari C. Symbolic Play in School-Aged Minimally Verbal Children with Autism Spectrum Disorder. J Autism Dev Disord. 2018 May;48(5):1436-1445. doi: 10.1007/s10803-017-3388-6. PMID 29170936
- [Result] Almirall D, DiStefano C, Chang YC, Shire S, Kaiser A, Lu X, Nahum-Shani I, Landa R, Mathy P, Kasari C. Longitudinal Effects of Adaptive Interventions With a Speech-Generating Device in Minimally Verbal Children With ASD. J Clin Child Adolesc Psychol. 2016 Jul-Aug;45(4):442-56. doi: 10.1080/15374416.2016.1138407. Epub 2016 Mar 8. PMID 26954267
- [Result] Kasari C, Kaiser A, Goods K, Nietfeld J, Mathy P, Landa R, Murphy S, Almirall D. Communication interventions for minimally verbal children with autism: a sequential multiple assignment randomized trial. J Am Acad Child Adolesc Psychiatry. 2014 Jun;53(6):635-46. doi: 10.1016/j.jaac.2014.01.019. Epub 2014 Mar 12. PMID 24839882
- [Result] Pizzano M, Shire S, Shih W, Levato L, Landa R, Lord C, Smith T, Kasari C. Profiles of minimally verbal autistic children: Illuminating the neglected end of the spectrum. Autism Res. 2024 Jun;17(6):1218-1229. doi: 10.1002/aur.3151. Epub 2024 May 27. PMID 38803132
- [Derived] Kasari C, Shire S, Shih W, Kaiser A, Lord C, Levato L, Smith T, Almirall D. Adaptive Intervention for School-Age, Minimally Verbal Children With Autism Spectrum Disorder in the Community: Primary Aim Results. J Am Acad Child Adolesc Psychiatry. 2025 Jun;64(6):674-685. doi: 10.1016/j.jaac.2024.10.020. Epub 2025 Jan 24. PMID 39864797